CLINICAL TRIAL: NCT02352844
Title: Phase II Study of Everolimus in Patients With Advanced Solid Malignancies With TSC1, TSC2, NF1, NF2, or STK11 Mutations
Brief Title: Everolimus in Patients With Advanced Solid Malignancies With TSC1, TSC2, NF1, NF2, or STK11 Mutations
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201502067
Record Dates: First submitted 2015-01-28; First posted 2015-02-02 (Estimated); Results first posted 2018-10-02 (Actual); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Solid Malignancy; Solid Tumor
MeSH Terms: interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm 1 (everolimus) (Experimental): Everolimus is an oral drug which will be administered on an outpatient basis at a dose of 10 mg daily on a 28-day cycle.
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: Everolimus
  Other Names: RAD001; Afinitor; Votubia

SUMMARY:
The purpose of this research study is to look at participants with solid tumor malignancies and specific mutations respond to treatment with everolimus.

DETAILED DESCRIPTION:
Cancer is a molecularly heterogeneous disease comprised of complex genomic alterations in common and overlapping pathways. Somatic inactivating mutations in tuberous sclerosis complex 1 (TSC1) gene were recently identified as potential markers of response to mTOR therapy. Everolimus is an oral derivative of rapamycin. At the cellular and molecular level, everolimus acts as a signal transduction inhibitor, and selectively inhibits mTOR. We hypothesize that everolimus will exhibit clinical activity in solid malignancies harboring TSC1, TSC2, NF1, NF2, or STK11 mutations.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of advanced (metastatic, recurrent, or unresectable) cancer with mutations in any of the following genes: TSC1, TSC2, NF1, NF2 or STK11.
* Must have failed at least 1 standard of care systemic therapy for their malignancy
* Measurable disease defined as lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as >10 mm with CT scan, as >20 mm by chest x-ray, or >10 mm with calipers by clinical exam.
* Prior therapy (chemotherapy, radiation therapy, and surgery) is allowed if completed at least 2 weeks prior to registration and if all treatment-related toxicities are resolved to ≤ CTCAE grade 1, with the exception of alopecia and hematologic values otherwise meeting the bone marrow function criteria specified below.
* At least 18 years of age.
* ECOG performance status ≤ 2
* Normal bone marrow and organ function as defined below:

  * Leukocytes > 3,000/mcL
  * Absolute neutrophil count > 1,500/mcL
  * Platelets > 100,000/mcL
  * Hemoglobin > 9.0 g/dL
  * Total serum bilirubin ≤ 2.0 x IULN
  * AST(SGOT)/ALT(SGPT) ≤ 2.5 x IULN (≤ 5.0 x IULN in patients with liver metastases)
  * Serum creatinine ≤ 1.5 x IULN OR creatinine clearance > 45 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
  * Fasting cholesterol ≤ 300 mg/dL OR ≤ 7.75 mmol/L AND fasting triglycerides ≤ 2.5 x IULN. NOTE: In case one or both of these thresholds are exceeded, the patient can only be included after initiation of appropriate lipid lowering medication
* Able to swallow tablets.
* Women of childbearing potential, defined as all women physiologically capable of becoming pregnant, must use highly effective methods of contraception during the study and for 8 weeks after. Women are considered post-menopausal and not of childbearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g., age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks prior to randomization. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow-up hormone level assessment is she considered not of childbearing potential.
* Male patients whose sexual partner(s) are women of childbearing potential must agree to use adequate contraception during the study and for 8 weeks after the end of treatment.
* Able to understand and willing to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable)

Exclusion Criteria:

* A history of other malignancy ≤ 3 years previous with the exception of basal cell or squamous cell carcinoma of the skin which were treated with local resection only or carcinoma in situ of the cervix.
* Taking an investigational agent within 4 weeks of initiation of everolimus.
* Symptomatic brain metastases. Known brain metastases are allowed if asymptomatic and previously treated.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to everolimus or other agents used in the study.
* Known impairment of GI function or GI disease that may significantly alter the absorption of oral everolimus.
* Currently taking CYP3A4 inhibitors or inducers (such as the antiepileptic drugs phenytoin, carbamazepine, or phenobarbital; cyclosporine; grapefruit or its juice; Seville oranges; starfruit; or St. John's wort)
* Chronic treatment with corticosteroids or other immunosuppressive agents. Topical or inhaled corticosteroids are allowed.
* Received live attenuated vaccine within 1 week of start of everolimus (i.e. intranasal influenza, measles, mumps, rubella, oral polio, BCG, yellow fever, varicella, and TY21a typhoid vaccines).
* Uncontrolled diabetes mellitus defined as HbA1c > 8% despite adequate therapy. Patients with a known history of impaired fasting glucose or diabetes mellitus may be included; however, blood glucose and antidiabetic treatment must be monitored closely throughout the trial and adjusted as necessary.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure of NYHA class III or IV, active coronary artery disease, unstable angina pectoris, cardiac arrhythmia, myocardia infraction ≤ 6 months prior to start of everolimus, uncontrolled hypertension (systolic pressure > 150 mmHg or diastolic pressure > 90 mmHg), uncontrolled seizure disorder, liver disease such as cirrhosis, decompensated liver disease, active and chronic hepatitis, known severely impaired lung function (spirometry and DLCO 50% or less of normal and 02 saturation 88% or less at rest on room air), active bleeding diathesis, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 14 days of study entry.
* Known HIV-positivity on combination antiretroviral therapy because of the potential for pharmacokinetic interactions with everolimus. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-10-07 (Actual); Primary Completion 2017-08-15 (Actual); Study Completion 2017-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Saiama Waqar, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to participant enrollment on 10/07/2015 and closed to participant enrollment on 06/28/2017.
Period: Overall Study
Arm/Group | Arm 1 (Everolimus)
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Arm 1 (Everolimus)
Number analyzed (Participants) | 12
Age, Continuous [Median (Full Range); unit: years] | 65 [40 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Response Rate (RR)
Description: The primary endpoint will be to describe the response rate using RECIST 1.1. Response rate will be defined as complete response (disappearance of all target lesion) plus partial response (a least a 30% decrease in the sum of diameters of target lesions).
Time Frame: Completion of treatment (estimated average of 6 months)
Population: 4 participants were not evaluable for this outcome measure as they discontinued treatment prior to disease assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 (Everolimus)
Number analyzed (Participants) | 8
Participants | 1

2. Secondary Outcome: Mutations Associated With Therapeutic Response
Description: -To correlate mutations in the mTOR pathway with therapeutic response with everolimus
Time Frame: Completion of treatment (estimated average of 6 months)
Population: 4 participants were not evaluable for this outcome measure as they discontinued treatment prior to disease assessment and are not evaluable for this outcome measure. Out of the 8 remaining participants, only one participant had a response (complete response to therapy) and specific mutations associated with response are described below.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 (Everolimus)
Number analyzed (Participants) | 1
Participants
  STK11 c.375-2del | 1
  STK11 c.375-8C>G | 1

3. Secondary Outcome: Genetic Changes Associated With Disease Progression
Description: -To investigate the genetic changes associated with disease progression following treatment with everolimus.
Time Frame: Completion of treatment (estimated average of 6 months)
Population: * Out of the 8 participants evaluable for response, only 6 were evaluable for this outcome measure because only 6 participants had disease progression
  * Please note that 1 participant had both NF1 c.7190C>T and NF1 c.7253C>T mutations in the sample
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 (Everolimus)
Number analyzed (Participants) | 6
Participants
  NF1 p.E8* | 1
  STK11 p.E199* | 1
  NF1 p.Y489C | 1
  STK11 exon 1 E33X | 1
  STK11 L282fs*5 | 1
  NF1 c.7190C>T | 1
  NF1 c.7253C>T | 1

ADVERSE EVENTS:
Time Frame: From start of treatment through 30 days after completion of treatment (estimated average of 7 months)
Arm/Group | Arm 1 (Everolimus)
All-Cause Mortality (participants affected / at risk) | 2/12
Serious Adverse Events (participants affected / at risk) | 8/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 (Everolimus) (N=12)
Abdominal pain (Gastrointestinal disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1
Biliary obstruction (Hepatobiliary disorders) | 1
Blood bilirubin increased (Investigations) | 1
Constipation (Gastrointestinal disorders) | 2
Death NOS (General disorders) | 1
Death due to progressive disease (General disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Flank Pain (Musculoskeletal and connective tissue disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Pericardial Effusion (Cardiac disorders) | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Portal vein thrombosis (Vascular disorders) | 1
Skin infection (Infections and infestations) | 1
Thromboembolic event (Vascular disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 (Everolimus) (N=12)
Activated partial thromboplastin time prolonged (Investigations) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Agitation (Psychiatric disorders) | 1
Alkaline phosphatase increased (Investigations) | 3
Anemia (Blood and lymphatic system disorders) | 5
Anorexia (Metabolism and nutrition disorders) | 3
Anxiety (Psychiatric disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Aspartate aminotransferase increased (Investigations) | 4
Atrial fibrillation (Cardiac disorders) | 2
Bruising (Injury, poisoning and procedural complications) | 1
Chills (General disorders) | 3
Confusion (Psychiatric disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Creatinine increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Depression (Psychiatric disorders) | 1
Diarrhea (Gastrointestinal disorders) | 4
Dizziness (Nervous system disorders) | 1
Dry eye (Eye disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Edema limbs (General disorders) | 2
Fatigue (General disorders) | 4
Fever (General disorders) | 2
Flashing lights (Eye disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 3
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypertension (Vascular disorders) | 5
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 3
Hypocalcemia (Metabolism and nutrition disorders) | 3
Hypokalemia (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 3
Insomnia (Psychiatric disorders) | 1
Itchy eyes (Eye disorders) | 1
Lymphocyte count decreased (Investigations) | 6
Mucositis oral (Gastrointestinal disorders) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Nail changes (Skin and subcutaneous tissue disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Nausea (Gastrointestinal disorders) | 1
Neutrophil count decreased (Investigations) | 2
Non-cardiac chest pain (General disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Pericardial Effusion (Cardiac disorders) | 2
Platelet count decreased (Investigations) | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Purpura (Skin and subcutaneous tissue disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 2
Rectal hemorrhage (Gastrointestinal disorders) | 1
Sweating (General disorders) | 1
Thromboembolic event (Vascular disorders) | 1
Trismus (Musculoskeletal and connective tissue disorders) | 1
Urinary frequency (Renal and urinary disorders) | 1
Vomiting (Gastrointestinal disorders) | 4
Weight loss (Investigations) | 1
White blood cell decreased (Investigations) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-15): https://cdn.clinicaltrials.gov/large-docs/44/NCT02352844/Prot_SAP_000.pdf